CLINICAL TRIAL: NCT03748355
Title: Using Pharmacogenetics to Identify Patients With Polypharmacy at Risk of Medication Adverse Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Simon Kung, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-006182
Record Dates: First submitted 2018-11-18; First posted 2018-11-20 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Psychiatric Disorder
Keywords: Polypharmacy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacogenetic Analysis (Other): A pharmacogenetic analysis will be completed for each participant upon inclusion into the study
  Interventions: Genetic: Pharmacogentic Analysis

INTERVENTIONS:
Genetic: Pharmacogentic Analysis — Participant will complete a buccal swab and it will be sent off to OneOme for analysis. When the results are available, the study investigators will review the medications for potential drug-drug and drug-genotype interactions. The risk for interactions will be classified as low, medium or high. The investigators will then communicate to the clinical team taking care of the patient these results and whether medication changes are recommended to minimize the drug-drug and drug-genotype interactions.
  Other Names: OneOme Pharmacogentic Analysis

SUMMARY:
The Researchers are trying to learn more about how individuals break down and process medications based on their genes. The Researchers want to find out whether subjects will have fewer side effects if they take different medications based on their pharmacogenomics profile.

DETAILED DESCRIPTION:
The Researchers are trying to learn more about how individuals break down and process medications based on their genes. The Researchers are doing this in order to assess the number of potential genotype-based drug interactions and side effects in patients with polypharmacy as well as to assess the number of potential individualized (based on the patient's genotype) drug interactions and side effects in these patients. After completing the OneOme genetic testing and relaying those results to the patients care team, the Researchers will then assess, at 30 days post-recommendations, whether the medication recommendations to reduce individualized drug interactions and adverse effects were followed, and (2) whether the adverse effects decrease compared to admission.

Patients will be recruited from the inpatient units listed in the inclusion criteria and, upon admission, each patient will complete a 24 item questionnaire measuring medication side effects, have a review of their medications for potential drug-drug and drug-genotype interactions (classified as low, medium or high risk), and then undergo the buccal swab to collect the DNA cells which will then be sent to OneOme for analysis. When the results are available, the study investigators will review the medications again for potential drug-drug and drug-genotype interactions and then communicate to the patients clinical team those results and whether medication changes are recommended to minimize the drug-drug and drug-genotype interactions.

Thirty days after the recommendations are communicated to the patient's clinical team, the patient will be contacted by phone. During this phone call, the following information will be obtained:

1. The patient's current medication list.
2. The patient's 24 item questionnaire measuring medication side effects.
3. The patient's one item self rating of improvement Once this phone call is completed, the research team will determine whether the medication recommendations were followed by the patient's clinical team, whether the adverse effects decreased compared to hospital admission, and whether the patient reported improvement.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* Hospitalized on Generose 2E (Acute Care Psychiatry), 3E (Medical and Geriatric Psychiatry), or 3W (Mood Disorders Unit).
* A voluntary patient
* Having 5 or more medications (scheduled or as needed) on their medication list.
* Ability to give informed consent

Exclusion Criteria:

* Patient with cognitive impairments such as moderate to severe dementia.
* Patients who do not communicate in English or cannot comprehend the rating scales used.
* Patients who have had pharmacogenetics testing performed within the previous 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-14 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

PRIMARY OUTCOMES:
Reduction of Potential Drug Interactions | 30 days
  Reduction of potential drug interactions risk measured by the numbers in low, medium and high categories.

SECONDARY OUTCOMES:
Reduction of Side Effects | 30 days
  Reduction of side effects as measured by side effects rating scale. Improvement of patient's self-assessment via the questionnaire item.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Kung, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials